CLINICAL TRIAL: NCT05650723
Title: Zanubrutinib and Venetoclax as Initial Therapy for CLL With Obinutuzumab Consolidation in Patients With Minimal Residual Disease Positivity (BruVenG)
Brief Title: Zanubrutinib and Venetoclax as Initial Therapy for Chronic Lymphocytic Leukemia (CLL) With Response-based Obinutuzumab
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: BeiGene (Industry); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 22-05024874
Record Dates: First submitted 2022-12-06; First posted 2022-12-14 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Leukemia, Lymphocytic, Chronic, B-Cell
Keywords: Chronic Lymphocytic Leukemia; CLL; Small Lymphocytic Lymphoma; SLL
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — zanubrutinib; venetoclax; obinutuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Double Therapy (Zanubrutinib plus Venetoclax) (Experimental): All participants will receive an initial 3 cycles of zanubrutinib monotherapy. This lead-in period will then be followed by 12 cycles of zanubrutinib and venetoclax combination therapy. All participants will complete 12 cycles of zanubrutinib and venetoclax combination therapy or 15 cycles of total treatment. Peripheral blood and bone marrow MRD assessments will occur at C16D1. Participants will continue on double combination treatment for an additional 1 month while results of MRD testing are obtained. In total, all participants will be on treatment for at least 16 full cycles. Participants that meet definition of MRD negativity will stop therapy at C17D1 and enter an observation phase with study visits every 3 months. Participants that remain MRD positive at C16D1 will enter the triple therapy (zanubrutinib, venetoclax, and obinutuzumab) arm.
  Interventions: Drug: Zanubrutinib Pill; Drug: Venetoclax Pill
- Triple Therapy (Zanubrutinib, Venetoclax, and Obinutuzumab) (Experimental): Participants that meet definition of MRD positivity at C16D1 will enter the triple therapy arm (zanubrutinib, venetoclax, and obinutuzumab). These participants will continue combination therapy with zanubrutinib and venetoclax, but will also receive 6 cycles of obinutuzumab starting at C17D1. In this subgroup, peripheral blood and bone marrow MRD assessments will occur after an additional 6 cycles of the triplet combination therapy (C23D1) at which point all participants will stop study treatment regardless of MRD status.
  Interventions: Drug: Zanubrutinib Pill; Drug: Venetoclax Pill; Drug: Obinutuzumab Injection

INTERVENTIONS:
Drug: Zanubrutinib Pill — 320 mg once per day by mouth
  Other Names: Brukinsa
Drug: Venetoclax Pill — 400 mg once per day by mouth following the standard ramp-up schedule (20mg daily PO week 1, 50mg daily PO week 2, 100mg daily PO week 3, 200mg daily PO week 4, followed by 400mg PO daily week 5)
  Other Names: Venclexta
Drug: Obinutuzumab Injection — 1000 mg IV given every 28 days
  Other Names: Gazyva
  Arms: Triple Therapy (Zanubrutinib, Venetoclax, and Obinutuzumab)

SUMMARY:
Bruton's tyrosine kinase inhibitors (BTKi), anti-CD20 antibodies, and the B cell lymphoma 2 inhibitor (BCL-2i) venetoclax are drug classes used to treat patients with chronic lymphocytic leukemia/small lymphocytic leukemia (CLL/SLL). Anti-CD20 therapy may not be required for all patients. The investigators hypothesis is that it may be better to give anti-CD20 therapy (obinutuzumab) only to patients that still have detectable cancer in their blood (minimal residual disease [MRD]) after being treated with a combination of two oral medications, zanubrutinib (a BTKi ) and venetoclax (a BCL-2i), instead of giving a combination of three drugs to all patients from the start of treatment. This strategy, if effective, will prevent overtreatment with anti-CD20 antibodies; reduce side effects of treatment while potentially increasing MRD negativity rates; and will possibly make the anti-CD20 antibody therapy more effective given the low tumor burden present when utilized. This study will test this hypothesis by treating subjects with 3 cycles of a zanubrutinib monotherapy lead-in, in order to debulk and mitigate tumor lysis risk, followed by 13 cycles of zanubrutinib and venetoclax combination therapy. Subjects who are both peripheral blood and bone marrow MRD negative at the completion of the 13 cycles of combination therapy will stop treatment and enter an observation phase every 3 months. Subjects that are MRD positive will continue combination therapy with zanubrutinib and venetoclax for an additional 6 cycles but also receive 6 cycles of obinutuzumab in order to augment response and increase MRD negative rates for the overall treated cohort.

DETAILED DESCRIPTION:
This is an open label, phase II, investigator-initiated clinical trial of 50 subjects. Subjects with CLL/SLL who have treatment indications per the 2018 International Workshop for CLL (iwCLL) will be eligible to enroll. The investigators hypothesize that anti-CD20 therapy may not be required for all patients and a response-adapted strategy will prevent over treatment of a significant number of patients and reduce toxicity of treatment while still achieving a high rate of MRD negativity. The investigators also hypothesize that late addition of anti-CD20 therapy can eliminate low burden residual disease in subjects and maximize undetectable MRD negativity in subjects who remain MRD positive.

All subjects will initiate induction therapy with 3 cycles of zanubrutinib monotherapy in order to debulk subjects and mitigate tumor lysis risk. This lead-in period will then be followed by 12 cycles of zanubrutinib and venetoclax combination. Standard ramp-up protocols for venetoclax based on TLS risk assessed prior to C4D1 will be utilized. All subjects will complete 12 cycles of zanubrutinib and venetoclax combination therapy or 15 cycles of total treatment. Peripheral blood and bone marrow MRD assessments will occur at C16D1. Subjects will continue on combination treatment for an additional 1 month while results of MRD testing are obtained. In total, all subjects will be on treatment for at least 16 full cycles. Subjects that meet definition of MRD negativity will stop therapy at C17D1 and enter an observation phase with study visits every 3 months. Subjects that meet definition of MRD positivity will continue combination therapy with zanubrutinib and venetoclax, but will also receive 6 cycles of obinutuzumab starting at C17D1. In this subgroup, peripheral blood and bone marrow MRD assessments will occur after an additional 6 cycles of the triplet combination therapy (C23D1) at which point all subjects will stop study treatment regardless of MRD status.

ELIGIBILITY:
Inclusion Criteria

1. Subject must be able to voluntarily sign and date an informed consent, approved by an Independent Ethics Committee (IEC)/Institutional Review Board (IRB), prior to the initiation of any screening or study specific procedures.
2. Subject must be ≥ 18 years of age.
3. Subject must have confirmed diagnosis of CLL/SLL based upon 2018 iwCLL Guidelines.

   a. Please note, participants with SLL must have identifiable B-cells in peripheral blood or bone marrow consistent with CLL/SLL immuno-phenotype, based on flow-cytometry, in order to be enrolled
4. Subject must have indications for treatment per the 2018 iwCLL Guidelines.
5. Subject has an Eastern Cooperative Oncology Group (ECOG) performance score of ≤ 2.
6. Subject must have adequate organ function defined as:

   1. Creatinine clearance ≥ 30 mL/min (as estimated by the Cockcroft-Gault equation or the Modification of Diet in Renal Disease equation, or as measured by nuclear medicine scan or 24-hour urine collection).
   2. Aspartate aminotransferase (AST)/serum glutamic oxaloacetic transaminase, and alanine aminotransferase (ALT)/serum glutamic pyruvic transaminase ≤ 2.5 × upper limit of normal (ULN) unless due to CLL/SLL.
   3. Serum total bilirubin < 3.0 × ULN (unless documented Gilbert's syndrome)
7. Subject must have adequate bone marrow function and meet the below thresholds unless approved by sponsor if cytopenias are felt to be due to significant marrow involvement of CLL:

   1. Absolute neutrophil count ≥ 1.0 x103/μL
   2. Hemoglobin ≥ 7 g/dL (can be transfused up to 1 week prior to study enrollment)
   3. Platelets ≥ 75,000 cells/μL OR platelets ≥ 30,000 cells/μL if clearly due to disease under study (per investigator discretion)
8. Subjects of childbearing potential must be willing to comply with pregnancy prevention interventions (as defined in Section 4.4)

Exclusion Criteria

A subject will be ineligible for the study if he/she meets the following criteria:

1. Previous exposure to any systemic anti-cancer therapy as a treatment for CLL/SLL, including but not limited to chemotherapy, immunotherapy, radiotherapy, hormone therapy (other than contraceptives, hormone-replacement therapy or megestrol acetate) or investigational therapy.
2. Subject with a history of malignancy except for non-melanoma skin cancers. Subjects treated with curative intent via methods of local resection and or locally targeted anticancer treatment and are free of malignancy for at least 35 years from treatment end will be allowed to enroll. Adjuvant hormonal therapy will be allowed at time of enrollment if the subject otherwise is not excluded by the 3-year waiting period.
3. Subject requires chronic immunosuppressive therapy for any reason or was treated with immunosuppressive therapy within 6 months of study entry.
4. Subjects with active autoimmune hemolytic anemia or immune thrombocytopenia purpura.
5. Subject with prolymphocytic leukemia or Richter's Transformation.
6. Active bleeding, or history of bleeding diathesis (e.g., hemophilia or von Willebrand disease).
7. Subject requires warfarin or equivalent vitamin K antagonist.
8. Uncontrolled or active significant infection requiring systemic treatment, subjects are eligible if they have completed antibiotic therapy 2 weeks prior to study enrollment.
9. History of suspected or confirmed PML
10. Clinically significant cardiovascular disease including the following:

    1. Myocardial infarction within 6 months before screening.
    2. Unstable angina within 3 months before screening.
    3. New York Heart Association class III or IV congestive heart failure
    4. History of clinically significant arrhythmias (eg, sustained ventricular tachycardia, ventricular fibrillation, torsades de pointes).
    5. QT interval corrected with Fridericia's formula (QTcF) > 480 milliseconds based on Fridericia's formula.
    6. History of Mobitz II second-degree or third-degree heart block without a permanent pacemaker in place.
    7. Uncontrolled hypertension as indicated by a minimum of 2 consecutive blood pressure measurements showing systolic blood pressure > 170 mmHg and diastolic blood pressure > 105 mmHg at screening.
11. Patients with stroke or CNS hemorrhage within 6 months.
12. Pregnant or breastfeeding.

14. Major surgical procedure within 28 days of first dose of study drug. If a subject had surgery, they must have recovered adequately from any toxicity or complications before the first dose of study drug.

15. Has difficulty with or is unable to swallow oral medication or has significant gastrointestinal disease that would limit absorption of oral medication.

16. Subject is known to be positive for human immunodeficiency virus (HIV). 17. Active hepatitis C, as confirmed by being positive for Hep C RNA by PCR. 18. Active hepatitis B infection documented by a positive PCR for Hep B DNA. If hepatitis B serology is positive for hepatitis B core antibody, but Hep B DNA PCR is negative, patient is eligible to enroll.

19. Subject requires:

1. Strong and moderate CYP3A inhibitors within 7 days prior to the initiation of study treatment.
2. Strong and moderate CYP3A inducers within 7 days prior to the initiation of study treatment.
3. Steroid therapy for anti-neoplastic intent with the exception of inhaled steroids for asthma, topical steroids, or replacement/stress corticosteroids within 7 days prior to the first dose of study drug administration.
4. Consumed grapefruit, grapefruit products, Seville oranges (including marmalade containing Seville oranges), or star fruit within 3 days prior to the first dose of study drug and throughout venetoclax administration.

   20. Known hypersensitivity reactions (e.g., anaphylaxis) to obinutuzumab or any of the excipients, including serum sickness with prior obinutuzumab use.

   21. Vaccination with live vaccine ≤28 days prior to start of treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-05-08 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of total patients that have achieved undetectable minimal residual disease (MRD) at cycle 16, as assessed via peripheral blood | Cycle 16 (Month 16)
  The primary endpoint of C16 peripheral blood MRD negativity at cycle 16 will be represented as a percentage of total patients. This will be calculated on both efficacy evaluable and intention to treat basis. These will be estimated with a 90% confidence interval using Clopper-Pearson method based on exact binomial distribution. A cycle is defined as 28 days.
Percentage of total patients that have achieved undetectable minimal residual disease (MRD) at cycle 16, as assessed via bone marrow aspirate | Cycle 16 (Month 23)
  The primary endpoint of C16 bone marrow MRD negativity at cycle 16 will be represented as a percentage of total patients. This will be calculated on both efficacy evaluable and intention to treat basis. These will be estimated with a 90% confidence interval using Clopper-Pearson method based on exact binomial distribution.
Percentage of eligible patients that have achieved undetectable minimal residual disease (MRD) at cycle 23, as assessed via peripheral blood | Cycle 23 (Month 23)
  The co-primary endpoint of C23 peripheral blood MRD negativity rate will be presented as a percentage of patients that achieve undetectable MRD at C23, who were found to be MRD positive at C16 and went on to receive at least one dose of obinutuzumab. This will be calculated on both efficacy evaluable and intention to treat basis. These will be estimated with a 90% confidence interval using Clopper-Pearson method based on exact binomial distribution.
Percentage of eligible patients that have achieved undetectable minimal residual disease (MRD) at cycle 23, as assessed via bone marrow aspirate | Cycle 23 (Month 23)
  The co-primary endpoint of C23 bone marrow MRD negativity rate will be presented as a percentage of patients that achieve undetectable MRD at C23, who were found to be MRD positive at C16 and went on to receive at least one dose of obinutuzumab. This will be calculated on both efficacy evaluable and intention to treat basis. These will be estimated with a 90% confidence interval using Clopper-Pearson method based on exact binomial distribution.

SECONDARY OUTCOMES:
Percentage of total participants who experience adverse events (AEs) through cycle 16 | Cycle 16 (Month 16)
  The secondary endpoints measuring toxicity will be tabulated using CTCAE 5.0. Numbers of participants experiencing adverse events (AEs) will be represented as a percentage through cycle 16.
Percentage of participants receiving triplet therapy who experience AEs through cycle 23 | Cycle 23 (Month 23)
  The secondary endpoints measuring toxicity will be tabulated using CTCAE 5.0. Participants who were MRD positive at cycle 16 and who receive obinutuzumab will have AEs tabulated as a percentage of total patients in the obinutuzumab consolidation phase of the study.
36-month Progression Free Survival (PFS) | 36 months
  Thirty-six-month PFS will be determined via Kaplan-Meier methods. PFS will be defined as the time from first treatment day until progression or death from any cause, as assessed at 36 months. Patients who do not experience an event or lost to follow-up will be censored.
36-month Overall Survival (OS) | 36 months
  36-month OS will be determined via Kaplan-Meier methods. OS will be defined as the time from first treatment day until death from any cause as assessed at 36-months. Patients who do not experience an event or lost to follow-up will be censored.
Percentage of patients treated with doublet therapy (zanubrutinib and venetoclax) that have achieved undetectable minimal residual disease (MRD) at 24-months, as assessed via peripheral blood | 24 months
  The percentage of patients who were treated with doublet therapy of zanubrutinib and venetoclax who achieve undetectable MRD at 24 months, as assessed with via peripheral blood, will be calculated on both efficacy evaluable and intention to treat basis. These will be estimated with a 90% confidence interval using Clopper-Pearson method based on exact binomial distribution. A cycle is defined as 28 days.
Percentage of patients treated with doublet therapy (zanubrutinib and venetoclax) that have achieved undetectable minimal residual disease (MRD) at 36-months, as assessed via peripheral blood | 36 months
  The percentage of patients who were treated with doublet therapy of zanubrutinib and venetoclax who achieve undetectable MRD at 36 months, as assessed with via peripheral blood, will be calculated on both efficacy evaluable and intention to treat basis. These will be estimated with a 90% confidence interval using Clopper-Pearson method based on exact binomial distribution. A cycle is defined as 28 days.
Percentage of patients treated with triplet therapy (zanubrutinib and venetoclax) that have achieved undetectable minimal residual disease (MRD) at 36-months, as assessed via peripheral blood | 36 months
  The percentage of patients who were treated with triplet therapy who achieve undetectable MRD at 36 months, as assessed with via peripheral blood, will be calculated on both efficacy evaluable and intention to treat basis. These will be estimated with a 90% confidence interval using Clopper-Pearson method based on exact binomial distribution. A cycle is defined as 28 days.
36-month Time to Next Treatment (TTNT) | 36 months
  36-month TTNT will be determined via Kaplan-Meier methods. TTNT will be measured from the start of treatment to the date of next line of treatment after stopping therapy. Obinutuzumab consolidation will not be considered a second line of treatment. Any treatment directed at CLL after stopping therapy will be considered a next therapy. Subjects will be followed prospectively and for 36 months from start of initial therapy to calculate a 3 year TTNT. Subjects that die will be censored at time of death.
Percentage Change in Tumor Lysis Syndrome (TLS) Risk Score From Baseline to Cycle 4 | Baseline; Cycle 4, Day 1 (Month 4)
  Tumor lysis risk of high, medium, or low will be collected at baseline/screening. After 3 cycles of zanubrutinib debulking, TLS risk will be reassessed prior to Cycle 4 day 1. Subjects will have their new assessment, high, medium, or low recorded. Change in TLS risk category will be reported in aggregate and as a percentage change after debulking.
Overall Response rate | 36 months
  Overall response rate including all categories of response will be tabulated and calculated as total percentage of patients achieving a specific response on an intention to treat basis.

CONTACTS AND LOCATIONS:
Overall Officials: John Allan, M.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine/NewYork-Presberteryian Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No